CLINICAL TRIAL: NCT02629952
Title: Metabolic Benefits of Drinking Blueberry Tea in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menzies Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Michelle Keske, Senior Research Fellow, Menzies Institute for Medical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H0014873
Record Dates: First submitted 2015-12-03; First posted 2015-12-15 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes
Keywords: glucose tolerance; type 2 diabetes; blueberry tea
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry Tea (Experimental): 3 cups of blueberry tea per day x 4 weeks
  Interventions: Other: Blueberry Tea
- No Treatment (No Intervention): No Treatment

INTERVENTIONS:
Other: Blueberry Tea — Blueberry Tea
  Arms: Blueberry Tea

SUMMARY:
Plant derived compounds, e.g. flavonoids from dark chocolate, green tea, or blueberries, show great potential as nutraceuticals for the treatment of various diseases such as type 2 diabetes (T2D). Flavonoids have been suggested to improve glucose metabolism, reduce blood lipids, reduce oxidative stress and improve vascular function. For these reasons we recently investigated the effects of daily consumption of locally produced blueberry tea and demonstrated that this could partially restore insulin sensitivity in an animal model. We propose to translate these findings to assess the efficacy of this nutraceutical as a new treatment for improving glucose tolerance in people with T2D.

DETAILED DESCRIPTION:
Current treatments for T2D are limited, have unwanted side effects, and lose effectiveness over time. There is a growing public interest in the use of complementary and alternative approaches for treating insulin resistance and T2D. Blueberries, blueberry leaves and cinnamon have each been reported to improve insulin sensitivity or insulin action. Blueberry Boost™ is a locally produced Blueberry Tea and is a proprietary blend of dried blueberries (37% wt/wt), blueberry leaves, raspberry leaves, spearmint leaves and cinnamon.

It is well established that improving glycemic control is important for managing insulin resistance and T2D and the associated vascular pathologies that directly contribute to end-organ damage (microvascular disease), hypertension and cardiovascular disease (stroke, heart attack and heart failure). We have recently demonstrated that a unique blueberry tea blend fully restores the vascular insulin sensitivity in muscle of the high-fat fed insulin-resistant rat model and is associated with substantial improvements in muscle glucose uptake and whole body insulin sensitivity. We propose to translate these findings to assess the efficacy of this nutraceutical as a new treatment for improving glucose tolerance in people with T2D.

Aim: Determine whether chronic consumption (4 weeks) of blueberry tea can improve metabolic and vascular health in people with and without T2D.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years.
* Normal to overweight (BMI 19-35 kg/m2).
* On lifestyle or metformin only diabetes treatment.
* Normotensive (seated brachial blood pressure <160/100 mmHg).
* No history of T2D (e.g. fasting plasma glucose <7.0mM); or with clinically diagnosed T2D on metformin or lifestyle intervention only (e.g. fasting plasma glucose ≥7.0mM, HbA1c).
* Willing to drink blueberry tea for 4 weeks (3 times per day with meals).

Exclusion Criteria:

* Age <18 yrs or >76 yrs
* Morbidly obese with a BMI ≥36 kg/m2
* Not on lifestyle and/or metformin only treatment for diabetes (e.g. insulin injections, sulphonylureas).
* History of myocardial infarction or stroke
* History of malignancy within past 5 years (except for non-melanoma skin cancers)
* Current smoker
* History of severe liver disease
* History of drug or alcohol abuse
* Elective major surgery during the course of the study
* Pregnancy/lactation
* Currently consuming (or have regularly consumed in the past 2 months) blueberry tea, or supplements containing blueberries, blueberry leaves, raspberry leaves, spearmint or cinnamon.
* Participation or intention to participate in another clinical research study during the study period.
* Not willing to consume blueberry tea for 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-11; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Glucose Tolerance after 4 weeks of drinking blueberry tea. | 4 weeks
  Oral glucose tolerance test (75g glucose) measured on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design). Blood glucose and plasma insulin levels measured at 0, 15, 30, 60, 90 and 120 min following consumption of glucose load.

SECONDARY OUTCOMES:
Improvement in Hemoglobin A1c (HbA1c) levels after 4 weeks of drinking blueberry tea. | 4 weeks.
  HbA1c levels measured on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).
Improvement in fasting Serum Lipid (cholesterol, HDL, LDL,triglycerides) levels after 4 weeks of drinking blueberry tea. | 4 weeks
  Fasting serum lipids (cholesterol, HDL, LDL,triglycerides) measured on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).
Improvement in fasting serum pro-inflammatory cytokine (IL-6, IL-1b, CRP, TNFa) levels after 4 weeks of drinking blueberry tea. | 4 weeks
  Fasting serum pro-inflammatory cytokines (IL-6, IL-1b, CRP, TNFa) assessed by ELISA will be measured on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).
Improvement in fasting serum albumin levels after 4 weeks of drinking blueberry tea.. | 4 weeks
  Fasting serum albumin levels measured on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).
Fasting serum electrolytes (Na, K, Cl, HCO3). | 4 weeks
  Fasting serum electrolytes (Na, K, Cl, HCO3) measured on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).
Improvement in Resting Blood Pressure (central and brachial blood pressure) after 4 weeks of drinking blueberry tea. | 4 weeks
  Blood Pressure (central and brachial blood pressure) will be measured by Mobil-O-Graph and assessed on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).
Improvement in resting Augmentation Index after 4 weeks of drinking blueberry tea. | 4 weeks
  Augmentation index will be measured by Mobil-O-Graph and assessed on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).
Improvement in large artery stiffness after 4 weeks of drinking blueberry tea. | 4 weeks
  Large artery stiffness will be measured by Mobil-O-Graph and assessed on 3 occasions: at baseline, after 4 weeks of drinking blueberry tea, and after 4 weeks of no treatment (randomized cross-over design).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Keske, PhD, Principal Investigator — Menzies Institute for Medical Research
Locations (1):
- Menzies Institute for Medical Research, Hobart, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeFuria J, Bennett G, Strissel KJ, Perfield JW 2nd, Milbury PE, Greenberg AS, Obin MS. Dietary blueberry attenuates whole-body insulin resistance in high fat-fed mice by reducing adipocyte death and its inflammatory sequelae. J Nutr. 2009 Aug;139(8):1510-6. doi: 10.3945/jn.109.105155. Epub 2009 Jun 10. PMID 19515743
- [Background] Martineau LC, Couture A, Spoor D, Benhaddou-Andaloussi A, Harris C, Meddah B, Leduc C, Burt A, Vuong T, Mai Le P, Prentki M, Bennett SA, Arnason JT, Haddad PS. Anti-diabetic properties of the Canadian lowbush blueberry Vaccinium angustifolium Ait. Phytomedicine. 2006 Nov;13(9-10):612-23. doi: 10.1016/j.phymed.2006.08.005. Epub 2006 Sep 18. PMID 16979328
- [Background] Stull AJ, Cash KC, Johnson WD, Champagne CM, Cefalu WT. Bioactives in blueberries improve insulin sensitivity in obese, insulin-resistant men and women. J Nutr. 2010 Oct;140(10):1764-8. doi: 10.3945/jn.110.125336. Epub 2010 Aug 19. PMID 20724487
- [Background] Couturier K, Batandier C, Awada M, Hininger-Favier I, Canini F, Anderson RA, Leverve X, Roussel AM. Cinnamon improves insulin sensitivity and alters the body composition in an animal model of the metabolic syndrome. Arch Biochem Biophys. 2010 Sep 1;501(1):158-61. doi: 10.1016/j.abb.2010.05.032. Epub 2010 May 31. PMID 20515642
- [Background] Qin B, Nagasaki M, Ren M, Bajotto G, Oshida Y, Sato Y. Cinnamon extract prevents the insulin resistance induced by a high-fructose diet. Horm Metab Res. 2004 Feb;36(2):119-25. doi: 10.1055/s-2004-814223. PMID 15002064